CLINICAL TRIAL: NCT06733519
Title: Evaluation of TH104 for Moderate to Severe Pruritus in Primary Biliary Cholangitis: a Double-blind, Randomized, Placebo-controlled, Phase 2a Study
Brief Title: TH104 for the Treatment of Pruritus in Primary Biliary Cholangitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tharimmune Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TH104-108
Record Dates: First submitted 2024-12-03; First posted 2024-12-13 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2024-12

CONDITIONS: Pruritus; Primary Biliary Cholangitis
MeSH Terms: conditions — Pruritus; Liver Cirrhosis, Biliary | interventions — nalmefene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Drug: Nalmefene
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nalmefene — Th-104 Nalmefene Mucoadhesive Buccal strip
  Arms: Treatment
Drug: Placebo — Matching placebo to TH-104
  Arms: Control

SUMMARY:
A phase 2a, multicenter, randomized, double-blind, placebo-controlled study of TH104 in primary biliary cholangitis (PBC) participants with moderate to severe pruritus.

DETAILED DESCRIPTION:
Following written informed consent, participants with PBC and pruritus will be screened to establish study eligibility. Eligible participants will participate in a one-week observation period for baseline recording, to train participants in the use of electronic PRO tools, and establish baseline itch scores. Another eligibility assessment will be done at the end of this observation period (i.e., at baseline [Day 0]) to ensure that no changes in eligibility have occurred and to confirm that the participant remains eligible. At the baseline visit, participants will be randomized to receive placebo or TH104 treatment. Block randomization will be used, in a 1:2 ratio of placebo:TH104. Treatment will start with a 1-week dose escalation period in which participants will be escalated from 2 mg/day to 4 mg/day TH104 or matching placebo. This will be followed by 2 weeks of treatment with 8 mg and then 3 weeks of 16 mg of TH104 or matching placebo. Following the end of treatment, participants will enter a two-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18 to 75 years, inclusive, at the time of signing the informed consent form.
2. Diagnosis of PBC, as demonstrated by the participant presenting with at least 2 of the following criteria at the Screening Visit:

   1. history of sustained increased alkaline phosphatase (ALP) levels first recognized at least 6 months prior to the Screening Visit
   2. positive antimitochondrial antibodies (AMA) titer (>1:40 titer on immunofluorescence or M2 positive by enzyme-linked immunosorbent assay [ELISA])
   3. PBC-specific antinuclear antibodies (antinuclear dot and nuclear rim positive)
   4. liver biopsy consistent with PBC Note: Participants with compensated cirrhosis will be eligible for enrollment only after the DSMB reviewed the safety and tolerability of TH104 in the first 10 non-cirrhotic participants.
3. Screening ALP value below 10 × upper limit of normal (ULN).
4. Participants taking the following drugs may be enrolled to the study, as long as they are on stable doses for > 12 weeks prior to the Screening Visit; Ursodeoxycholic acid (UDCA) Obeticholic acid Elafibranor Seladelpar Fibrates such as bezafibrate and fenofibrate Cholestyramine Antihistamines
5. Symptoms of pruritus - rated as NRS > 4 for worst daily score:

   * At screening AND
   * At least on 4 days during the 1-week baseline observation period.
6. A woman is eligible to participate if she is not breast-feeding or pregnant, as confirmed by a negative serum human chorionic gonadotrophin (hCG) test or at least one of the following conditions applies:

   1. Non-reproductive potential defined as pre-menopausal with a documented tubal ligation or hysterectomy; or post-menopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 mIU/mL and estradiol <40 pg/mL (<147 pmol/L) is confirmatory]. Women on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods along with either a second form of highly effective contraception or barrier protection (condoms with spermicide) if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment;
   2. Reproductive potential and agrees to follow one of the contraception options methods for the specified duration of time.

   For men participating in the study and having a female partner - birth control methods described above will have to be used throughout the study.
7. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. Screening total bilirubin >2.0 x ULN.
2. Screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >4 x ULN.
3. Screening serum creatinine >2.5 mg/dL (221 µmol/L).
4. History or presence of hepatic decompensation (e.g., variceal bleeds, encephalopathy, or poorly controlled ascites).
5. History or presence of other concomitant liver diseases including hepatitis due to hepatitis B or C virus (HCV, HBV) infection, primary sclerosing cholangitis (PSC), alcoholic liver disease, definite autoimmune hepatitis or biopsy-proven non-alcoholic steatohepatitis (NASH/MASH/MAFLD).
6. Thyroid stimulating hormone (TSH) out of normal ranges.
7. Administration of the following drugs at any time during the 3 months prior to the Screening Visit: colchicine, methotrexate, azathioprine, opioids, opioids antagonists, or systemic corticosteroids.
8. Current or chronic history of inflammatory bowel disease, chronic diarrhea, Crohn's disease, or diarrhea related to malabsorption syndromes.
9. Based on averaged corrected QT interval (QTc) values of triplicate electrocardiograms (ECGs) obtained at least 5 minutes apart: QTc ≥450 msec; or QTc ≥480 msec in participants with Bundle Branch Block.
10. History of sensitivity to any of the study medications (or components thereof) or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
11. History of regular alcohol consumption within 6 months of the Screening Visit defined as an average weekly intake of >21 units for men or >14 units for women. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
12. A positive screening drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids, and benzodiazepines.
13. Where participation in the study would result in blood in blood sampling in excess of 500 mL within a 56-day period.
14. Treatment with sertraline and/or rifampicin < 4 weeks prior to the Screening Visit.
15. Clinically significant abnormality of the buccal mucosa which could impact drug absorption.
16. Participation in a clinical trial with an investigational product within 30 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer) before the first dosing in this study.
17. Decompensated liver disease (encephalopathy, ascites, or Child Pugh score > 10 points). Participants with compensated cirrhosis will be eligible for enrollment after the DSMB reviewed the safety and tolerability of TH104 for the first 10 non-cirrhotic participants).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to investigate the safety and tolerability of repeat doses of TH104 | 42 days
  Percentage of participants with treatment-related adverse events as coded by MedDRA.

SECONDARY OUTCOMES:
Difference in daily itch score between TH104 and placebo | 42 days
Change in participants reported outcome for PBC-40 questionnaire | 42 days
  The PBC-40 is a disease specific questionnaire that assess PBC related symptoms . The six domains of PBC-40 relate to fatigue, emotional, social, and cognitive function, general symptoms, and itch
Change in participants reported outcome for 5-D itch questionnaire. | 42 days
  The 5-D itch scale was developed as a brief but multidimensional questionnaire designed to be useful as an outcome measure in clinical trials. The five dimensions are degree, duration, direction, disability and distribution.
Change in participants reported outcome for EQ5D quality of life questionnaire | 42 days
  EQ-5D assesses health status in terms of five dimensions of health.
Change in Fatigue Severity Scale from baseline to the end of treatment. | 42 days
  The FSS questionnaire contains nine statements that rate the severity of fatigue symptoms

IPD SHARING:
Plan to Share IPD: Undecided